CLINICAL TRIAL: NCT01288248
Title: The Risk of Laryngospasm in Children is Similar to the Use of the Laryngeal Mask and the Endotracheal Tube in Children 2 Years to 14 Years: Clinical Trial Randomized Noninferiority
Brief Title: Noninferiority Clinical Trial With Laryngeal Mask and Endotracheal Tube
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Olga Luci-a Giraldo Salazar, MD, Anestesiologist, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anestudea-001
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Laryngospasm; Bradycardia
Keywords: Airway; Airway laryngeal mask; Endotracheal tube; Respiration artificial; Laryngospasm; Safety of airway laryngeal mask
MeSH Terms: conditions — Laryngismus; Bradycardia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Airway laryngeal mask classic (Experimental): Ventilation with Airway laryngeal mask classic during surgery
  Interventions: Device: Airway laryngeal mask classic
- endotracheal tube (Active Comparator): Ventilation with endotracheal tube during surgery
  Interventions: Device: endotracheal tube

INTERVENTIONS:
Device: Airway laryngeal mask classic — This group includes patients with the randomization process are assigned to use Classic laryngeal mask as a method to secure the airway after induction of anesthesia, which will be maintained during surgery and removed the patient asleep once you are done the surgical procedure to determine the presence or absence of laryngospasm.
  The laryngeal mask mark to be used will laryngeal Mask Device ® which comes in different sizes and sterilized in ethylene oxide. The size of the Classic laryngeal mask is used according to the weight assigned
  Other Names: airway laryngeal mask proseal
  Arms: Airway laryngeal mask classic
Device: endotracheal tube — This group includes patients with the randomization process are allocated to use endotracheal tube method for securing the airway after induction of anesthesia, which will be maintained during surgery and removed in the awake patient when you finish the surgical procedure to determine the presence or absence of laryngospasm.
  The marks of the endotracheal tube will be one of the following: Kendall Curity ®, Well Lead Medical ®, Meditec ®, which are not reusable. The size of the endotracheal tube be allocated according to age.
  Other Names: laryngeal tube
  Arms: endotracheal tube

SUMMARY:
The purpose of this study is to determine whether the use of laryngeal mask classic as method for securing the airway in the population of 2 years to 14 years is associated with risk of laryngospasm as compared with the use of endotracheal tube.

DETAILED DESCRIPTION:
Laryngospasm, defined as closure of the glottis as a protective reflex secondary to abnormal stimulation (7), with a reported incidence in the general population of 8.7 per 1000 patients undergoing surgical procedures (8), is considered the most common event among the complications in the management of pediatric airway, causing 40% of obstructive events after extubation (7-8), with incidents reported in the American pediatric population from 0.4% to 14% (8-9) for population under 6 years and 3.6% in > 6 years. Among the risk factors associated with the development of laryngospasm and anesthesia in children are: age, ASA (4), upper respiratory infection (10), among others, however in recent years has gained interest and generated dispute the association between this outcome and the type of device used to secure the airway during anesthesia. Although the endotracheal tube device is considered the "gold standard" for airway management, this has been associated with an increased incidence of laryngospasm (8), explained this phenomenon, apparently by direct stimulation because the tube into the larynx and trachea, which triggers, in theory, a posterior laryngeal reflex intense (11).

In recent years, with the advent of new devices for securing the airway, especially supraglottic use type Classic Laryngeal Mask (LM), it was thought that the main trigger of laryngospasm, laryngeal and tracheal stimulation caused by the endotracheal tube (ETT), would be resolved and will decrease the incidence of complications in the pediatric population; however, three recent prospective studies (10-11-12) is no statistically significant difference in incidence of laryngospasm among laryngeal mask and endotracheal tube. By contrast, two retrospective studies (6.4) have shown increased incidence of laryngospasm compared to ETT in children. In 2002, one of the aforementioned prospective studies (11), found an incidence of laryngospasm 11.2% versus 16.9% for ETT versus ML, respectively, but without an increase in relative risk statistically significant when comparing the ML to ETT.

In view of these findings and considering that most studies in this respect seem to have technical and methodological limitations, our objective is to determine by controlled clinical trial non inferiority the risk of laryngospasm with the endotracheal tube vs a device supraglottic, Classic Laryngeal Mask type as a method of airway patency in the pediatric population, assuming that the risk of laryngospasm with both devices is equal.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and III children, 1-14 years of age
* Children scheduled for surgery or therapeutic procedures under general anesthesia and fasting as defined in the fasting guidelines
* Responsible adult patients whose accept and sign the informed consent of study

Exclusion Criteria:

* Surgery of the head, neck, chest and/or abdomen (except the abdominal wall)
* Position different than the supine in surgery
* Malformations or anatomic abnormalities of the face and airway
* Procedures over 3 hours
* Patients with pulmonary aspiration risk: morbid obesity, intestinal obstruction, gastrointestinal bleeding, gastroparesis, gastroesophageal reflux
* Patients with limited mouth opening or cervical spine extension and classified as difficult airway

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 338 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Laryngospasm clinically manifested as inspiratory stridor and/or expiratory, no breath sounds, paradoxical movement of the thorax and abdomen and desaturation, bradycardia, central cyanosis. | The appearance of the outcome will be measured from anesthetic induction until the patient is fully awake
  It should be noted that once the subject of study presents the primary outcome may end up changing the device to improve ventilation.

SECONDARY OUTCOMES:
Desaturation defined as SaO2 < 90% in pulse oximetry associated with laryngospasm | from anesthetic induction until the patient is fully awake
Presence of bradycardia in the cardioscope as reported for the age. | from anesthetic induction until the patient is fully awake

CONTACTS AND LOCATIONS:
Overall Officials: Olga Lucia Giraldo Salazar, MD, MsH, Principal Investigator — Foundation Hospital San Vicente de Paul, St. Vincent Foundation
Locations (1):
- Hospital Foundation St. Vincent de Paul, Medellín, Antioquia, Colombia